CLINICAL TRIAL: NCT02659410
Title: Studying the Impact of Thermal Stress (Heat) Representative of Occupational Settings on Pulmonary Absorption and Toxicokinetics of 3 Organic Solvents
Brief Title: Impact of Thermal Stress on Pulmonary Absorption and Toxicokinetics of 3 Organic Solvents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Montréal (Other)
Collaborators: Institut de Recherche Robert-Sauvé en Santé et en Sécurité du Travail (Other)
Responsible Party: Principal Investigator, Sami Haddad, Professor, Université de Montréal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14-140-CERES-P; 2013-0012 (Other Grant/Funding Number: IRSST)
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Heat
Keywords: Physiologically based pharmacokinetic modeling; Organic solvents
MeSH Terms: interventions — Heat-Shock Response; 3',5'-dichloromethotrexate; Administration, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Heat stress (Experimental): 4h exposure to heat stress alone or in combination with different solvents. Solvent concentrations are equal to their TLV. Heat conditions are 21, 25 and 30°C (WBGT). Inhalation exposure for all solvents and demal exposure for toluene.
  Interventions: Other: Heat stress (21); Other: Heat stress (25); Other: Heat stress (30); Other: Heat Stress (21) +TOL; Other: Heat stress (25) + TOL; Other: Heat stress (21) + TOL; Other: Heat stress (21) + ACE; Other: Heat stress (25) + ACE; Other: Heat stress (30) + ACE; Other: Heat stress (21) + DCM; Other: Heat stress (25) + DCM; Other: Heat stress (30) + DCM; Other: Heat stress (21) + TOL (dermal); Other: Heat stress (25) + TOL (dermal); Other: Heat stress (30) + TOL (dermal)

INTERVENTIONS:
Other: Heat stress (21) — 4h exposure to heat (WBGT of 21°C), no solvent
Other: Heat stress (25) — 4h exposure to heat (WBGT of 25°C), no solvent
Other: Heat stress (30) — 4h exposure to heat (WBGT of 30°C), no solvent
Other: Heat Stress (21) +TOL — 4h exposure to heat (WBGT of 21°C) + Toluene (concentration = TLV)
Other: Heat stress (25) + TOL — 4h exposure to heat (WBGT of 25°C) + Toluene (concentration = TLV)
Other: Heat stress (21) + TOL — 4h exposure to heat (WBGT of 30°C) + Toluene (concentration = TLV)
Other: Heat stress (21) + ACE — 4h exposure to heat (WBGT of 21°C) + Acetone (concentration = TLV)
Other: Heat stress (25) + ACE — 4h exposure to heat (WBGT of 25°C) + Acetone (concentration = TLV)
Other: Heat stress (30) + ACE — 4h exposure to heat (WBGT of 30°C) + Acetone (concentration = TLV)
Other: Heat stress (21) + DCM — 4h exposure to heat (WBGT of 21°C) + Dichloromethane (concentration = TLV)
Other: Heat stress (25) + DCM — 4h exposure to heat (WBGT of 25°C) + Dichloromethane (concentration = TLV)
Other: Heat stress (30) + DCM — 4h exposure to heat (WBGT of 30°C) + Dichloromethane (concentration = TLV)
Other: Heat stress (21) + TOL (dermal) — 4h exposure to heat (WBGT of 21°C) + Toluene (concentration = TLV), participants breath normal air through a mask for evaluation of dermal absorption.
Other: Heat stress (25) + TOL (dermal) — 4h exposure to heat (WBGT of 25°C) + Toluene (concentration = TLV), participants breath normal air through a mask for evaluation of dermal absorption.
Other: Heat stress (30) + TOL (dermal) — 4h exposure to heat (WBGT of 30°C) + Toluene (concentration = TLV), participants breath normal air through a mask for evaluation of dermal absorption.

SUMMARY:
In Quebec, thousands of workers are concomitantly exposed to heat and chemical compounds. Exposure to heat induces physiological responses that help maintaining a stable body temperature. Those changes can affect organ functions implicated in absorption and metabolism. According to literature, those changes could lead to increased concentrations of chemical compounds in the body and their toxicity. Therefore, the aim of this study is to evaluate the pulmonary absorption and toxicokinetics of 3 organic solvents in heat stress conditions in volunteers exposed in a inhalation chamber. Results will then be used to develop PBPK models that will allow to predict organic solvent kinetics when coexposed with heat.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18,5 et 25 kg/m3

Exclusion Criteria:

* Smoking
* Respiratory, cardiovascular and neurological problems
* History of exposure to solvents
* Chronic medication
* Abusive and/or chronic alcohol consumption
* Alcohol consumption 24h before or 18h following exposure

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-08 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Respiratory rate | 4hour
  Respiratory rate will be monitored continuously for 4hour with a respirometer
Cardiac frequency | 4hour
  Cardiac frequency will be monitored continuously for 4hour with a respirometer
Minute ventilation | 4hour
  Minute ventilation will be monitored continuously for 4hour with a respirometer
Tidal volume | 4hour
  Tidal volume will be monitored continuously for 4hour with a respirometer
Solvent in blood | 4,5hour
  Solvents concentrations will be measured in blood samples collected at different times (t=0, 2, 4 and 4.5hour).
Solvent or metabolite in urine | 18hour
  Solvent or metabolite concentrations (o-cresol for toluene exposures) will be measured for urine samples collected at different times (t=0, 4, 10 and 18hour).
Solvent in exhaled air | 6hour
  Solvents concentrations will be measured in exhaled air samples collected at different times (t=0, 1.5, 3, 4.5 and 6hour).

SECONDARY OUTCOMES:
Oxygen consumption | 4hour
  oxygen consumption will be monitored continuously for 4hour with a respirometer
Carbonic dioxide production | 4hour
  carbonic dioxide production will be monitored continuously for 4hour with a respirometer
Body temperature | 4hour
  Body temperature is monitored continuously by telemetry

CONTACTS AND LOCATIONS:
Overall Officials: Sami Haddad, Ph.D, Study Director — Université de Montréal
Locations (1):
- Université de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Marchand A, Menard J, Brochu P, Haddad S. Modeling the impact of heat stress on the toxicokinetics of toluene and acetone. Arch Toxicol. 2024 Feb;98(2):471-479. doi: 10.1007/s00204-023-03646-6. Epub 2023 Dec 21. PMID 38127129